CLINICAL TRIAL: NCT04517929
Title: Effectiveness of Group Psychotherapy in Patients With Fibromyalgia Syndrome, Randomized Controlled Study
Brief Title: Effectiveness of Group Psychotherapy in Patients With Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Meryem Burcu Turkoglu, Principal invastigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-6.1T/49
Record Dates: First submitted 2020-07-27; First posted 2020-08-19 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Fibromyalgia Syndrome
Keywords: fibromyalgia; group therapy; group psychotherapy; pain; depression; anxiety
MeSH Terms: conditions — Fibromyalgia; Pain; Depression; Anxiety Disorders | interventions — Psychotherapy, Group

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Patients in this group will receive recommendations regarding lifestyle change, exercise, and nutrition related to fibromyalgia.
- intervention group (Experimental): Patients in this group will receive recommendations regarding lifestyle change, exercise, and nutrition related to fibromyalgia and group psychotherapy.
  Interventions: Other: Group Psychotherapy

INTERVENTIONS:
Other: Group Psychotherapy — 9 week group psychotherapy, given by a psychologist trained in group psychotherapy.
  Arms: intervention group

SUMMARY:
The hypothesis of the study is that group therapy in fibromyalgia patients can provide significant improvement in pain, fatigue, anxiety and depression levels and emotional expressions.

DETAILED DESCRIPTION:
The purpose of our study; to determine the effectiveness of group psychotherapy in the treatment of Fibromyalgia Syndrome.

Patients who received 9 weeks of group therapy and those who did not, at the beginning of treatment, at the end of 9 weeks and 6 months after treatment will be evaluated using The Short Form-36, Fibromyalgia Impact Questionnaire, Revised Fibromyalgia Impact Questionnaire, Hospital Anxiety and Depression Scale, Fatigue Severity Scale, Beck Depression Inventory, Beck Anxiety Inventory, Pain Beliefs Scale, Emotional Expression Questionnaire, Visual Analogue Scale, Childhood Trauma Questionnaire, 2016 Fibromyalgia Diagnostic Criteria.

At the end of the study, individuals are expected to show less depressive symptoms and anxiety symptoms compared to the beginning of the study, and it is thought that their complaints about pain will decrease.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia Syndrome diagnosed according to 2016 Fibromyalgia Syndrome diagnostic criteria
* Volunteers between the ages of 18-65
* Literate volunteers
* Volunteering to participate in group work
* There is no obstacle to attend the sessions regularly every week

Exclusion Criteria:

* Who cannot participate in 9-week group therapy
* Under 18, over 65 years old
* Confused enough to not be able to complete and understand the scales given cognitively
* Having serious mental illness (eg Psychotic disorder, Mental Retardation etc.)
* Illiterate individuals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain-Visual Analog Scale | At the beginnning of the study ,through study completion-8th week, after study completion -6th month
  Chronic musculoskeletal pain in Fibromyalgia syndrome patients, in this scale minumum value is 0, maximum value is 10, higher scores means worse outcome.
Change in Depression-Beck Depression Inventory | At the beginnning of the study ,through study completion-8th week, after study completion -6th month
  Depression in Fibromyalgia patients
Change in Anxiety-Beck Anxiety Inventory | At the beginnning of the study ,through study completion-8th week, after study completion -6th month
  Anxiety in Fibromyalgia patients

SECONDARY OUTCOMES:
Change in The Short Form (36) Health Survey | At the beginnning of the study ,through study completion-8th week, after study completion -6th month
  The Short Form (36) Health Survey
Change in Fibromyalgia Impact Questionaire | At the beginnning of the study ,through study completion-8th week, after study completion -6th month
  Fibromyalgia Impact Questionaire
Change in Revised Fibromyalgia Impact Questionnaire | At the beginnning of the study ,through study completion-8th week, after study completion -6th month
  Revised Fibromyalgia Impact Questionnaire
Change in Hospital Anxiety and Depression Scale | At the beginnning of the study ,through study completion-8th week, after study completion -6th month
  Hospital Anxiety and Depression Scale, in this scale minumum value is 0, maximum value is 21, high scores mean worse outcome.
Change in The Fatigue Severity Scale | At the beginnning of the study ,through study completion-8th week, after study completion -6th month
  The Fatigue Severity Scale, In this scale consisting of 9 items, each item is scored between 1 and 7 (1 = strongly disagree, 7 = totally agree) and the total score is calculated by taking the average of 9 items, high scores mean worse outcome.
Change in Pain beliefs questionnaire | At the beginnning of the study ,through study completion-8th week, after study completion -6th month
  Pain beliefs questionnaire
Change in Emotional Expression Questionnaire | At the beginnning of the study ,through study completion-8th week, after study completion -6th month
  Emotional Expression Questionnaire
CHILDHOOD TRAUMA QUESTIONNAIRE | At the beginning of the study
  CHILDHOOD TRAUMA QUESTIONNAIRE
Change in 2016 Fibromyalgia Syndrome Criteria | At the beginnning of the study ,through study completion-8th week, after study completion -6th month
  2016 Fibromyalgia Syndrome Criteria
  2016 Fibromyalgia Diagnostic Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Simin HEPGULER, Prof, Study Chair — Ege University; Basak DURDU AKGUN, Dr, Principal Investigator — Ege University; Ece Cinar, Assistant Prof, Principal Investigator — Ege University
Locations (1):
- Ege University Faculty of Medicine, Izmır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clauw DJ, Arnold LM, McCarberg BH; FibroCollaborative. The science of fibromyalgia. Mayo Clin Proc. 2011 Sep;86(9):907-11. doi: 10.4065/mcp.2011.0206. PMID 21878603
- [Background] Jones GT, Atzeni F, Beasley M, Fluss E, Sarzi-Puttini P, Macfarlane GJ. The prevalence of fibromyalgia in the general population: a comparison of the American College of Rheumatology 1990, 2010, and modified 2010 classification criteria. Arthritis Rheumatol. 2015 Feb;67(2):568-75. doi: 10.1002/art.38905. PMID 25323744
- [Background] Bennett RM, Jones J, Turk DC, Russell IJ, Matallana L. An internet survey of 2,596 people with fibromyalgia. BMC Musculoskelet Disord. 2007 Mar 9;8:27. doi: 10.1186/1471-2474-8-27. PMID 17349056
- [Background] Arnold LM, Hudson JI, Keck PE, Auchenbach MB, Javaras KN, Hess EV. Comorbidity of fibromyalgia and psychiatric disorders. J Clin Psychiatry. 2006 Aug;67(8):1219-25. doi: 10.4088/jcp.v67n0807. PMID 16965199
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Hisli N. Beck Depresyon Ölçeği'nin bir Türk örnekleminde geçerlik ve güvenirliği. Psikoloji Dergisi 1988; 6:118-122.
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Ulusoy M, Şahin NH, Erkmen H. Turkish version of the Beck Anxiety Inventory: Psychometric properties. J Cognit Psychother 1996; 12:163- 172
- [Background] Edwards LC, Pearce SA, Turner-Stokes L, Jones A. The Pain Beliefs Questionnaire: an investigation of beliefs in the causes and consequences of pain. Pain. 1992 Dec;51(3):267-272. doi: 10.1016/0304-3959(92)90209-T. PMID 1491853
- [Background] Bernstein DP, Fink L, Handelsman L, Foote J, Lovejoy M, Wenzel K, Sapareto E, Ruggiero J. Initial reliability and validity of a new retrospective measure of child abuse and neglect. Am J Psychiatry. 1994 Aug;151(8):1132-6. doi: 10.1176/ajp.151.8.1132. PMID 8037246
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092
- [Background] Kuzucu Y. , "Duyguları İfade Etme Ölçeği'nin Uyarlanması: Geçerlik Ve Güvenirlik Çalışmaları" Kastamonu Eğitim Dergisi, Cilt:19 No:3, 2011,779-792.